CLINICAL TRIAL: NCT06923397
Title: Interrupting Sedentary Time to Improve Cardiometabolic Health and Toxicity in Patients With Lymphoma Receiving Chemotherapy: The iSTAND Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-765
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Lymphoma, Hodgkin; Lymphoma, Non-Hodgkin; Sedentary Behavior
Keywords: Lymphoma; Hodgkin Lymphoma; Lymphoma, Hodgkin; Lymphoma, Non-Hodgkin; Non-Hodgkin Lymphoma; Sedentary Behavior
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrupted Sedentary Time Intervention (Experimental): The first 3 participants enrolled with be placed into the intervention group. After this, participants will be randomized in a group allocation ratio of 2:1 using permuted blocked design with varying block size and stratified by treatment plan. 14 participants will complete:
  * Baseline visit
  * Standard of care chemotherapy treatment regimen
  * Daily exercise sessions in-clinic up to 4x weekly and at home 6 days per week
  * Week 14 post-intervention visit
  Interventions: Behavioral: Interrupted Sedentary Time Intervention
- Usual Care Control Group (No Intervention): Participants will be randomized in a group allocation ratio of 2:1 using permuted blocked design with varying block size and stratified by treatment plan. 7 participants will complete:
  * Baseline visit
  * Standard of Care chemotherapy treatment regimen
  * Week 14 visit
  * Participants will be offered Fitbit activity tracker and resistance bands at the end of the study.

INTERVENTIONS:
Behavioral: Interrupted Sedentary Time Intervention — A 12-week, semi-supervised exercise intervention comprised of reminder prompts, counseling, and activities of walking, cycling, and resistance band exercise for at-home and in-clinic settings. Supervision will be under an exercise trainer. Resistance bands, Libre Pro continuous blood sugar monitor, and Fitbit and ActivPAL trackers will be provided to participants.
  Arms: Interrupted Sedentary Time Intervention

SUMMARY:
This study aims to see if a 12-week exercise program designed to reduce long periods of inactivity is feasible in newly diagnosed lymphoma participants receiving R-CHOP or POLA-R-CHP chemotherapy treatments, and whether it can improve heart health and reduce chemotherapy drug side effects.

DETAILED DESCRIPTION:
The purpose of this study is to see if a 12-week exercise program designed to reduce long periods of inactivity is feasible in newly diagnosed lymphoma participants receiving R-CHOP or POLA-R-CHP chemotherapy treatments, and whether it can improve heart health and reduce chemotherapy drug side effects.

Participants will be randomized into one of two groups: Group A: Interrupted Sedentary Time Intervention vs. Group B: Usual Care Control Group. Randomized means a participant is placed into a study group by chance.

The research study procedures include screening for eligibility, assessments of fitness and physical health, blood tests, and questionnaires.

Participation in this research study is expected to last about 3 months.

It is expected that about 24 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign informed consent prior to any study- related procedures.
* Patients diagnosed with lymphoma.
* Will receive first line R-CHOP or POLA-R-CHP chemotherapy regimens, patients do not need to be within a certain timeframe from diagnosis.
* Aged ≥18 years; due to the rarity of the disease in those <18 years, this age bracket will not be included.
* Engaging in ≤60-minutes of structured moderate or vigorous intensity exercise.
* Have physician clearance to participate in exercise.
* Speak English.
* Willing to travel to Dana-Farber Cancer Institute for necessary data collection and exercise sessions.
* Access to a phone that can receive text messages.

Exclusion Criteria:

* Unstable comorbidities that prevent participation in moderate-to-vigorous intensity exercise. Patients with unstable comorbidities likely require supervised exercise for safety, and part of this study involves unsupervised exercise; therefore, for safety reasons, these persons are excluded.
* Participate in more than 60 minutes of structured moderate-to-vigorous exercise per week over the last month. Excess additional exercise is a confounding factor in assessing the effect of the current interrupted sedentary time intervention.
* Patients receiving treatment for other active malignancies (except basal cell carcinoma). This study is exclusively targeting lymphoma chemotherapy-related effects.
* Subjects who in the opinion of the investigators may not be able to comply with the safety monitoring requirements of the study.
* Unable to travel to DFCI Longwood campus for necessary data collection and chemotherapy infusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention Completion Rate (Feasibility) | 12 weeks
  Intervention feasibility is defined as: 1) A participant completes ≥70% of the supervised activity breaks on at least 3 out of the 4 infusion appointments. 2) A participant completes ≥70% of the prescribed home-based resistance activity breaks on at least 48 days out of the possible 68 days (12 week) intervention (excluding the 4 infusion days and 1 rest day per week) (i.e., meet interrupting sedentary behavior goals across at least 70% of the intervention). 3) A participant completes ≥70% of the prescribed home-based step goals (i.e., >250 steps per hour) on at least 48 days out of the possible 68 days (12 week) intervention (excluding the 4 infusion days and 1 rest day per week) (i.e., meet interrupting sedentary behavior goals across at least 70% of the intervention).
Refusal Rate | 12 weeks
  Defined as ≤50% of eligible screened participants refuse to complete intervention.
Retention Rate | 13 weeks
  Retention of consented participants to study end is ≥70%.
Acceptability of Intervention Measure (AIM) Scale | 13 weeks
  Assessed by the Acceptability of the Intervention Measures, a 4-item measure rated on a 5-point Likert scale with answers ranging from "Completely disagree" to "Completely agree." A total scores range is 4 to 20 with a higher score indicating greater acceptability. The intervention will be deemed acceptable by participants if ≥70% of participants have a mean score ≥ 4 on the AIM.
Acceptability Exit Survey | 13 weeks
  The intervention will be deemed acceptable by participants if 1) ≥70% of participants report "agree" or "strongly agree" to the prompt "Participation in this study helped me reduce my daily sedentary time" and 2) ≥70% of participants report "probably" or "yes" to the prompt "I would recommend this program to other patients being treated for cancer."

SECONDARY OUTCOMES:
Participant Glucose Level | Assessed for one week at each timepoint (baseline & post-intervention).
  Glucose levels will be assessed by constant glucose monitoring where an average of >180 mg/dl will be considered hyperglycemic.
Participant Insulin Resistance | Assessed for one week at each timepoint (baseline & post-intervention).
  Insulin resistance will be assessed by calculating Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) from fasting blood samples where values >1.9 will be considered insulin resistant.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu